CLINICAL TRIAL: NCT07212660
Title: A Multi-center, Randomized-controlled, 12-month, Split-mouth, Non-inferiority Clinical Trial to Compare the Safety and Performance of Two Different Curing Modes in the Direct Filling Therapy With a Flowable Bulk Fill Composite in Class I and II Deciduous Teeth
Brief Title: A Clinical Trial to Compare the Safety and Performance of Two Different Curing Modes in the Direct Filling Therapy in Deciduous Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTCS 369512033
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries; Insufficient Dental Filling
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Split-mouth design: each patient receives 2 dental fillings (test and control treatment in the same patient)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast curing mode (Experimental): Composite restoration is cured with Turbo mode (5 seconds with 2000 mW/cm²).
  Interventions: Device: Fast curing mode
- Conventional curing mode (Other): Composite restoration is cured with High mode (10 seconds with 1200 mW/cm²).
  Interventions: Device: Conventional curing mode

INTERVENTIONS:
Device: Fast curing mode — Composite restoration is cured with Turbo mode (5 seconds with 2000 mW/cm²).
  Arms: Fast curing mode
Device: Conventional curing mode — Composite restoration is cured with High mode (10 seconds with 1200 mW/cm²).
  Arms: Conventional curing mode

SUMMARY:
The overall aim of this clinical investigation is to assess the clinical performance and safety of composite restorations cured with fast curing mode (5 seconds with 2000 mW/cm²) in primary molars.

DETAILED DESCRIPTION:
Dental interventions in young children are challenging due to limited compliance and anxiety. Moisture control during the placement of resin composite fillings is particularly difficult, as children need to remain calm. Reducing treatment time benefits both children and dentists.

The planned clinical investigation aims to evaluate the clinical performance and safety of posterior restorations on primary teeth using a flowable composite with a fast curing mode (5 seconds, 2000 mW/cm²) compared to a conventional curing mode (10 seconds, 1200 mW/cm²).

ELIGIBILITY:
Inclusion Criteria:

* Consent of a legal representative (usually parents)
* 2 deciduous molars in the need of direct filling therapy class I and/or II in different quadrants (primary or secondary caries, filling loss)
* Classification of caries: caries of all sizes in deciduous molars are included unless they can be treated with fissure sealing (ICDAS 3, 4, 5)
* Sufficient language skills of legal representative and children
* Teeth in the need of indirect pulp capping if necessary (Operator decision)

Exclusion Criteria:

* Cognitive impairment not age-appropriate
* Sensitive tooth (pain at night, irritation-persistent pain, buccal swelling, percussion sensitivity)
* Teeth with severely resorbed roots (anormal tooth mobility)
* Direct pulp capping
* Pulpotomy of an adjacent tooth in the same appointment
* Noncompliant child
* Allergies to material or anaesthetics used in the study
* Sufficient isolation not possible

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 4-10 days after placement of the dental fillings
  The assessment of postoperative pain will be done by using the Wong-Baker Faces Pain rating Scale and includes questions about type and duration of pain, intensity of pain and the type of stimulus causing the pain. Values of 0 and 2 in the Wong-Baker Faces Pain Rating Scale are considered as no pain and values >2 as pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - N|DENT Zahnarztpraxis, Herzogenbuchsee, Canton of Bern
  - Zahnarztpraxis Chrüzhof, Willisau, Canton of Lucerne

IPD SHARING:
Plan to Share IPD: No